CLINICAL TRIAL: NCT07237477
Title: Comparison of the Site Effect Model Prediction and BIS Predicted by Eleveld for Propofol in Slow and Rapid Inductions
Brief Title: Reevaluation Prediction of the Effect Site Propofol Eleveld Model Using Slow and Fast Induction
Acronym: fast or slow E
Status: Completed | Type: Observational
Sponsor: Pablo O. Sepulveda (Other)
Responsible Party: Sponsor-Investigator, Pablo O. Sepulveda, Dr. Med., Universidad del Desarrollo
Organization: Universidad del Desarrollo (Other)
Other Study IDs: Hospital Base San José Osoro
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia for Elective Surgery Patients; Anesthesia Brain Monitor; Pharmacodynamics
Keywords: Propofol, Eleveld model, induction flow, CONOX,
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: the prediction of the Eleveld propofol model in effect site mode TCI induction: Patients ASA 1-2, 18 to 70 years, will be induced using propofol TCI in effect site mode EC60 of the Eleveld PKPD model and compared with the EEG CONOX behavior, If lost of responsiveness (LOR) was not reached, we climb up 0,5 ug/ml every 3 min. At LOR calculated effect site concentration will be used as reference to mantain anesthesia level.
  Interventions: Drug: Evaluation of the prediction of from the propofol PKPD model including in TCI pumps using fast (Effect site mode TCI) or slow (plasma TCI mode) induction
- Group 2: the prediction of the Eleveld propofol model in TCI plasma mode: Patients ASA1-2, 18-70 years, scheduled for elective surgery longer than 1 hour. Induced with TCI plasma mode using the Eleveld PKPD model. The infusion will begin using a target plasma of 3 ug/ml, and scale every 3 minutes in 0,5 ug/ml until Loss of responsiveness (LOR). At LOR the calculated effect site concentration will be used as reference to mantain anesthesia level. EEG (CONOX or BIS) will be used to evaluate the prediction of the model.
  Interventions: Drug: Evaluation of the prediction of from the propofol PKPD model including in TCI pumps using fast (Effect site mode TCI) or slow (plasma TCI mode) induction

INTERVENTIONS:
Drug: Evaluation of the prediction of from the propofol PKPD model including in TCI pumps using fast (Effect site mode TCI) or slow (plasma TCI mode) induction — Using TCI technology and EEG monitoring (CONOX) we will induce loss of responsiveness using the fast induction (Group 1) or slow induction (Group 2) and compare the prediction of the effect site model (PD) in each type of induction.

SUMMARY:
Patients ASA1-2, 18 to 70 years old, scheduled for elective surgery with personal conset to participate, will be randomised into two groups using different induction mode. TCI effect site mode induction or TCI plasma mode induction both using the Elevelt PKPD propofol model. Standard monitoring (EKG, SaO2, PCo2et, NIAP), and Conox/ and or BIS EEG monitor to evaluate the prediction.

The model's prediction will be compared with values provided by the Conox/BIS index for both groups and between them. The study will be conducted during the 20 minutes after Loss of responsiveness.

DETAILED DESCRIPTION:
Patients aged 18 to 70 years will be included. Patients allergic to propofol are excluded. Eleveld's PKPD model for propofol includes covariates for adjustment in administration with target-controlled infusion pumps. Induction to the site of effect will be performed using EC60 for each age, while slow induction will use the target plasma modality, starting at a target of 3 ug/ml and increasing by 0.5 ug/ml every 3 minutes until loss of consciousness. This is defined as the loss of response to voice and shoulder tap. The 20 minutes following loss of consciousness will be evaluated.

Biometric and gender characteristics of both groups, concomitant pathologies, and surgical times will be compared.

The temporal evolution of the propofol effect site predicted by the Eleveld model will be compared between the two types of induction using EEG (CONOX or BIS). To obtain the EEG index prediction by Eleveld it will be use the Tiva trainer software 2.0, simulating the evolution of the kinetics and effect site calculated by Eleveld in the infudion TCI pumps.

It is estimated that 20 patients per group are required to find a 20% difference in predicted versus actual EEG index with 90% power.

Statistical methods:

1. Data analysis tool: Stata 10 software
2. Statistics

   * Summary: Mean (central tendency) and standard deviation (dispersion)
   * Association: Student's t-test for continuous quantitative variables and Fisher's exact test for dichotomous variables.

ELIGIBILITY:
Inclusion Criteria: patients ASA 1-2 scheduled for elective surgery, Exclusion Criteria: patients with psychiatric disorders, allergic to propofol, not giving their consent to participate

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ASA1-2, 18-70 years, scheduled for elective surgery longer than 1 hour
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Prediction of the efect site propofol Eleveld model | The data will be retrieved directly from the infusion pumps and EEGs up to 20 minutes after the loss of clinical consciousness.
  The comparison betwen predicted and actual CONOX/BIS index will be made in two scenario: TCI effect site mode induction versus TCI plasma mode induction

CONTACTS AND LOCATIONS:
Overall Officials: José Gonzalez Gonzalez, PHD, Study Director — Departamento de Investigación Hospital osorno
Locations (1):
- Hospital Base san José de Osorno, Osorno, Los Lagos Region, Chile

IPD SHARING:
Plan to Share IPD: Yes
Part of the analysis will be conducted by Matthias Kreuzer Techische Universität München
Supporting Information: SAP
Time Frame: from 3 November 2025 to March 2026
Access Criteria: EEG data and concentration data calculated for each patient will be shared in individual folders via Google Drive.
URL: https://drive.google.com/drive

REFERENCES:
- [Result] Coetzee E, Coetzee JF, Haasbroek M. Predictive pharmacodynamic performance of the Eleveld pharmacokinetic-pharmacodynamic model for propofol: comparison of predicted and measured bispectral index. Br J Anaesth. 2024 Oct;133(4):785-792. doi: 10.1016/j.bja.2024.06.041. Epub 2024 Aug 23. PMID 39179443
- See also: this study discuss about the problem of the Eleveld effect site prediction using diferent induction flows — https://www.elsevier.es/es-buscar?cmbBuscador=00349356&txtBuscador=+Influence++of++rate++of++administration++on++the++mechanism++behind++propofol++induced++loss++of++consciousness